CLINICAL TRIAL: NCT05588817
Title: Expression of IRAK1 Gene rs1059703-related Single- Nucleotide Polymorphisms in Egyptian Patient With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa atef Abdelsalam, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh_Med_22_10_15
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Normal control
  Interventions: Genetic: PCR polymorphism
- Group 2 (Active Comparator): Diagnosed Rhomatoid arthritis patients
  Interventions: Genetic: PCR polymorphism

INTERVENTIONS:
Genetic: PCR polymorphism — PCR polymorphism in Rhomatoid arthritis patients in Egypt

SUMMARY:
Rheumatoid arthritis (RA) is known as a long-lasting inflammatory autoimmune disease affecting the diarthrodial joints, which is diagnosed by inflammation and hyperplasia in synovium, generation of RF and anti-citrullinated protein antibody (ACPA), deformity of cartilage and bone, systemic injuries involving cardiovascular, pulmonary, psychological, and skeletal disorders (McInnes and Schett., 2011).

ELIGIBILITY:
Inclusion Criteria:

* approval to sign an informed written consent, patient diagnosed rheumatoid arthritis, patient age range 17-85 year and both sexes are included.

Exclusion Criteria:

* Refusal to sign an informed written consent and patient with other autoimmune disease.

Ages: 17 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
rs1059703 PCR polymorphism in rhomatoid arthritis patients | 1 year
  PCR polymorphism

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes